CLINICAL TRIAL: NCT00596141
Title: Pilot Study to Evaluate the Use of OroScience Topical Oral Wound Emulsion in Post Operative Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OroScience, Inc. (Industry)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORO_PG_LSU_1_08
Record Dates: First submitted 2008-01-05; First posted 2008-01-16 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Oral Surgical Procedures; Pain
Keywords: oral periodontal gingival intraoral mucosal mucoperiosteal; Surgery, Oral
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conventional postoperative care and instructions on dental hygiene will be provided along with the TOWE treatment which consists of the patient dispensing TOWE into a disposable dental tray and placing the dental tray over the dental arch and covering the surgical site 3 times daily for a period of 7 days. At three (3) days and seven (7) days postoperatively, photographs will be taken of all vertical releasing incisions (before suture removal).
  Interventions: Device: OroScience Topical Oral Wound Emulsion
- 2 (No Intervention): Conventional postoperative care and instructions on dental hygiene.

INTERVENTIONS:
Device: OroScience Topical Oral Wound Emulsion — TOWE will be applied 3 times daily for a period of 7 days by the patient dispensing TOWE into a disposable dental tray and placing the dental tray over the dental arch and covering the surgical site.
  Arms: 1

SUMMARY:
The purpose of this pilot study is to determine if Topical Oral Wound Emulsion (TOWE) assists with dental wound healing and relieves pain from oral wounds.

ELIGIBILITY:
Inclusion Criteria:

* Planned dental treatment includes intraoral surgery involving full thickness mucoperiosteal flaps with at least one vertical releasing incision

Exclusion Criteria:

* Complicated medical history
* History of poor patient compliance
* Presence or placement of materials beneath the suture site

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Visible signs of inflammation scored on a scale of 1 to 4 by three (3) blinded investigators. | Three (3) and seven (7) days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Billie G Jeansonne, DDS, PhD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- LSU School of Dentistry, Dental Clinics, New Orleans, Louisiana, United States